CLINICAL TRIAL: NCT03461497
Title: Value-Based Care in Abdominal Surgery: Measuring Recovery Outcomes That Matter to Patients
Brief Title: Development of a Patient-Reported Outcome Measure to Assess Recovery After Abdominal Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Hospital São Paulo, Brazil (Unknown); Hokkaido University Hospital (Other); San Raffaele University Hospital, Italy (Other); Cleveland Clinic Florida (Other); The Cleveland Clinic (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Julio F Fiore Jr, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: VT 57203
Record Dates: First submitted 2018-03-02; First posted 2018-03-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Surgery
Keywords: Patient-Reported Outcome; Patient Outcome Assessment; Questionnaire; Self-Report; Abdominal Surgery; Postoperative Period; Recovery of Function; Psychometrics; Qualitative Research; Patient-Centered

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Cohort: Patients undergoing abdominal surgery

SUMMARY:
As surgery enters the era of value-based care, it is advocated that postoperative recovery be measured using patient-reported outcomes (PROs) as they provide a mean to incorporate the patient's perspectives and experiences into research and clinical decision-making. In abdominal surgery, this is currently precluded by the lack of PRO measures specifically developed and validated in the context of postoperative recovery.

The core goal of this research project is to develop a PRO measure aimed to assess postoperative recovery from the perspective of patients undergoing abdominal surgery. This project complies with the US Food and Drug Administration (FDA) and International Society for Pharmacoeconomics and Outcomes Research (ISPOR) guidelines for PRO development and will be conducted in three phases:

Phase 1: Qualitative interviews with patients to develop a conceptual framework and generate relevant items.

Phase 2: Use of Rasch Analysis for item-reduction and scale formation.

Phase 3: Further assessment of measurement properties based on traditional psychometric methods.

DETAILED DESCRIPTION:
OBJECTIVE:

To develop a comprehensive, conceptually relevant and psychometrically sound PRO measure to assess recovery after abdominal surgery.

OUTLINE:

* Phase 1(Conceptual framework and item generation): Semi-structured interviews focusing on patient lived experiences after abdominal surgery will be conducted to derive the "final conceptual framework of recovery after abdominal surgery". The interviews are guided by the "hypothesized conceptual framework" which is based on previous literature and expert input. This phase has a minimal targeted sample of 30 patients. To account for potential cross-cultural differences in recovery experiences, the study is enrolling patients from 4 international sites: McGill University Health Centre (Montreal, Canada), Hospital Sao Paulo (Sao Paulo, Brazil), Vita-Salute San Raffaele Hospital (Milan, Italy), and Hokkaido University Hospital (Sapporo, Japan). Interview audio recordings are transcribed, translated if required, and coded according to ICF (International Classification of Functioning, Disability and Health) domains. Codes for which saturation is reached will comprise the final conceptual framework of recovery. Items reflecting the essence of each domain will be generated and patient understanding of the items will be assessed through cognitive interviews. Items for which no problems have been identified and those successfully revised will be compiled into an item pool to be 'calibrated' in subsequent stages of PRO development.
* Phase 2 (Item selection and scoring- Rasch Analysis): In phase 2, the preliminary item pool generated in phase 1 will undergo refinement using Rasch Measurement Theory (RMT). Based on this analysis, items will be modified or eliminated to ensure that the novel PRO measure fits a linear continuum and produces meaningful scores. A target sample of 100 patients undergoing abdominal surgery will be recruited from three tertiary hospitals in Canada. The participants will complete the preliminary PRO measure at five time points: preoperatively, and on postoperative days (PODs) 1, 7, 30, and 90. Items that fail to fit the Rasch model will be revised or removed.
* Phase 3 (Validation using traditional psychometric methods): Further evaluation of the measurement properties of the novel PRO measure will be conducted using traditional psychometric methods. A total of 600 patients undergoing abdominal surgery will be recruited in five tertiary hospitals in Canada and in the United States. Participants will complete the PRO measure in different timepoints: preoperatively, and on PODs 1-7, 28, 60, and 90. Assessment of psychometric properties will focus on internal consistency, test-retest reliability, measurement error, hypothesis testing construct validity, responsiveness, and criterion validity. Interpretability will be assessed by estimating the minimal important difference (MID) using anchor-based methods.

ELIGIBILITY:
The following applies to all phases of the project.

Inclusion Criteria:

* Age ≥18 years old
* Abdominal surgery within three days to three months before enrolment
* Fluent in the local language
* Willing and able to provide written informed consent

Exclusion Criteria:

* Documented mental impairment
* Palliative care
* Advanced musculoskeletal, neurological, pulmonary or cardiac disorders
* Organ transplantation
* Cesarean section

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient's that have undergone abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome Measure (PRO) | 3 years
  PRO measure of recovery after abdominal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Julio F Fiore Jr, PhD, Principal Investigator — McGill University, Department of Surgery; Liane S Feldman, MD, Principal Investigator — McGill University, Department of Surgery
Locations (7):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic (Main Campus), Cleveland, Ohio
- Hospital São Paulo, São Paulo, Brazil
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal
- San Raffaele Hospital, Milan, Italy
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fiore JF Jr, Figueiredo S, Balvardi S, Lee L, Nauche B, Landry T, Mayo NE, Feldman LS. How Do We Value Postoperative Recovery?: A Systematic Review of the Measurement Properties of Patient-reported Outcomes After Abdominal Surgery. Ann Surg. 2018 Apr;267(4):656-669. doi: 10.1097/SLA.0000000000002415. PMID 28767559
- [Background] Alam R, Figueiredo SM, Balvardi S, Nauche B, Landry T, Lee L, Mayo NE, Feldman LS, Fiore JF Jr. Development of a patient-reported outcome measure of recovery after abdominal surgery: a hypothesized conceptual framework. Surg Endosc. 2018 Dec;32(12):4874-4885. doi: 10.1007/s00464-018-6242-9. Epub 2018 May 17. PMID 29777351
- [Background] Alam R, Montanez J, Law S, Lee L, Pecorelli N, Watanabe Y, Chiavegato LD, Falconi M, Hirano S, Mayo NE, Feldman LS, Fiore JF Jr. Development of a conceptual framework of recovery after abdominal surgery. Surg Endosc. 2020 Jun;34(6):2665-2674. doi: 10.1007/s00464-019-07044-x. Epub 2019 Aug 1. PMID 31372888
- [Background] Rajabiyazdi F, Alam R, Pal A, Montanez J, Law S, Pecorelli N, Watanabe Y, Chiavegato LD, Falconi M, Hirano S, Mayo NE, Lee L, Feldman LS, Fiore JF Jr. Understanding the Meaning of Recovery to Patients Undergoing Abdominal Surgery. JAMA Surg. 2021 Aug 1;156(8):758-765. doi: 10.1001/jamasurg.2021.1557. PMID 33978692